CLINICAL TRIAL: NCT01581164
Title: Studies of the Immune Response to Vaccination After Hematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: UCSF Protocol No. 112526
Record Dates: First submitted 2012-04-16; First posted 2012-04-20 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: blood; hematopoietic; stem; cell; transplant; vaccine; vaccination; recovery; immune; system
MeSH Terms: interventions — Influenza Vaccines; Chickenpox Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum will be collected and stored for immunologic analysis after vaccination. Samples will be cryopreserved. No cell lines will be created using samples procured on this protocol.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HSCT patients: Patients who have been treated with HSCT
  Interventions: Biological: Influenza vaccine; Biological: Varicella vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Influenza vaccine: Injection, post transplant
  Other Names: flu vaccine
Biological: Varicella vaccine — Varicella vaccine: Injection, post transplant
  Other Names: chicken pox vaccine

SUMMARY:
The purpose of this research study is to perform a serial analysis of immune function using blood cells and sera obtained from patients after vaccination following hematopoietic stem cell transplantation (HSCT). The focus of this study will be to characterize several immune parameters during the clinical course of HSCT and correlate these findings with the effect of vaccination.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation therapy is potentially curative for many malignant and non-malignant hematopoietic disorders. Disease recurrence and infection remain major causes of morbidity and mortality following HSCT. While innate immunity (myeloid and NK cell) is restored relatively quickly following HSCT, a prolonged period of lymphopenia occurs in all patients. This delay in lymphoid reconstitution is exacerbated with age and results in severely dampened adaptive immune responses. In children who have received chemotherapy and HSCT, T cell function generally recovers within 6 to twelve months. In contrast, lymphoid deficiency in adults may require years, and often never recovers to pre-transplant levels. Much of the delay in lymphocyte recovery is thought to be due to decreased thymic T cell production and export and the resulting expansion of treatment resistant T cell clones. Peripheral expansion of T cells in a lymphopenic setting leads to a narrowing of the TCR repertoire and manifests as a decrease in the magnitude of response to new antigens.

These long-lasting T cell deficiencies have been shown to play a direct role in post-transplant complications. There are many studies that correlate decreased T cell number and function (specifically CD4+ T cells) with an increase in post-transplant infections and relapse has been shown to be inversely proportional to T cell reconstitution following both autologous and allogeneic HSCT. Furthermore, this prolonged deficit in T cell function decreases the effectiveness of vaccination against tumour antigens and infectious diseases as well as other post-transplant immunotherapeutic strategies. Following HSCT, patients lose immunological memory not only to infectious microorganisms to which they were previously exposed but also bacterial and viral vaccines given prior to the HSCT , increasing the chance of infection post-transplant. Primary immunization requires antigenic stimulation and functionally mature T cells and therefore at least partial reconstitution of the T and B cell pools is necessary before successful reimmunization can occur.

This study presents an opportunity to analyze, at a systems level, the responses to vaccination in patients who are treated with HSCT. The expected high frequency of low responders to vaccination will permit comparisons of gene expression and immune cell activation between high and low responders as measured by the rate of seroconversion and HAI titers. The evaluation of live VZV vaccination is essential for these objective as the investigators hypothesize that live vaccination will induce a more specific immune response than dead (ie: influenza) vaccination. This study may also generate novel hypotheses about the mechanistic basis for reduced responses to vaccines post HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been treated with HSCT.
* Patients must be 5-70 years of age.
* For patients participating in Objective 3: Patients must be immunocompetent (no active GVHD and must be off all immunosuppression)

Exclusion Criteria:

* Patients who do not wish to participate or unable to provide the necessary blood samples required for the protocol.
* Patients with history of allergic reaction to a vaccination.
* Patient has had Guillain-Barre syndrome.
* Patients who are pregnant or become pregnant.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been treated with HSCT
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Immune response at Day 90 post vaccination. | Participants will have blood drawn at baseline and on Days 1, 7, 10, 28, and 90 post vaccinations following hematopoietic stem cell transplantation. Average study participation is 1-3 years post transplant.
  Participants will have blood drawn at baseline to Day 90 post vaccinations following hematopoietic stem cell transplantation. Average study participation is 1-3 years post transplant.

SECONDARY OUTCOMES:
Immune response | Participants will have blood drawn at 1 month intervals post hematopoietic stem cell transplantation . Average study participation is 1-3 years post transplant.
Immune response | Blood will drawn at baseline and Days 1, 7, 10, 28, and 90 post vaccination. Participants will receive the vaccine, 12-28 months post hematopoietic stem cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Venstrom, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States